CLINICAL TRIAL: NCT07233447
Title: Prevalence of H. Pylori in Stomach Cancers in the West Indies
Acronym: PyloCaGe
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de la Guadeloupe (Other)
Responsible Party: Sponsor
Other Study IDs: PAP_RIPH2_2020/27
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Oncology Epidemiology; Risk Factors
Keywords: H. Pylori; Guadeloupe; stomach cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The biological samples (serum, DNA, tumor) will be processed and stored for future research.
  The collection will be used for future somatic genetic analyses aimed at identifying additional disease-related risk factors. No analyses of constitutional (germline) genetic characteristics will be performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The incidence and mortality of stomach cancer are higher in the French West Indies than in mainland France. The prevalence of H. pylori infection associated with this cancer remains unknown in these populations. The main objective of the study is to estimate the prevalence of H. Pylori detected by immunohistochemistry in patients newly diagnosed with cancer.

DETAILED DESCRIPTION:
Stomach cancer is the 4th most common cancer site in the world and the 3rd cause of mortality. It is associated with infection by the Helicobacter Pylori bacterium, which colonizes the gastric mucosa in 80% of cases. The decrease of the prevalence of H. pylori infection in developed countries with the advent of antibiotic treatments is responsible for the decrease in the incidence of stomach cancer. But in the French West Indies, stomach cancer remains in excess incidence and mortality compared to France. The prevalence of H. pylori infection remains unknown, both in general population and in patients with stomach cancer. Eating habits combining high consumption of salt, meat and smoked fish could partly explain these high incidences. Furthermore, recent observations suggest that environmental risk factors (pesticides pollution) could also be involved in the occurrence of this cancer. Estimating the prevalence of H. pylori in stomach cancers will improve the epidemiological knowledge of this cancer with high incidence rates and prevention measures.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age residing in Guadeloupe for more than 6 months and with a primary diagnosis of gastric cancer
* Patient having read the information note and having signed the consent to participate in the study
* Patient with social security coverage.

Exclusion Criteria:

* Refusal to participate.
* Patient who could not answer the questionnaires
* Patient not affiliated to a social security scheme
* Patient under legal protection (judicial safeguard, guardianship, curatorship, etc.)
* Pregnant or breastfeeding woman
* Subject participating in another research study that includes an exclusion period still ongoing at the time of pre-inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients living in Guadeloupe for more than 6 months, referred to the gastroenterology departments of the University Hospital of Guadeloupe (CHUG) and to the gastroenterology practice of Dr. Durand, with an endoscopic diagnosis of gastric cancer confirmed by histopathological examination in one of the three endoscopy centers (CHUG, Polyclinique de la Guadeloupe, and Clinique des Eaux Claires), will be invited to participate in the study following their disclosure consultation.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2027-02-24 (Estimated); Study Completion 2027-02-24 (Estimated)

PRIMARY OUTCOMES:
detection of H. Pylori in immunohistochemistry | Baseline
  Detection of Helicobacter pylori will be performed by immunohistochemistry (IHC) on gastric biopsy samples collected at inclusion. The procedure aims to identify the presence of H. pylori antigens within the gastric mucosa using specific antibodies. The test will be conducted in a certified pathology laboratory according to standard diagnostic protocols. Results will be reported as positive or negative for H. pylori infection.

SECONDARY OUTCOMES:
positivity of anti H. Hylori serology by Elisa test | Baseline
  Positivity of anti-Helicobacter pylori serology determined by ELISA test performed on serum samples collected at inclusion. Results will be reported as positive or negative for H. pylori antibodies.

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Deloumeaux, MD PhD, Study Director — CHU de la Guadeloupe; Moana GELU-SIMEON, MD PhD, Study Chair — CHU de la Guadeloupe
Locations (2):
- Guadeloupe (2):
  - Cabinet Galeries de Houelbourg, Baie-Mahault
  - CHU de la Guadeloupe, Pointe-à-Pitre

IPD SHARING:
Plan to Share IPD: No